CLINICAL TRIAL: NCT02539797
Title: Improving Cognition in Schizophrenia Using Transcranial Direct Current Stimulation
Brief Title: Improving Cognition in Schizophrenia Using tDCS
Acronym: ICDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Yuri Rassovsky, Associate Research Psychologist, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 22017
Record Dates: First submitted 2015-08-26; First posted 2015-09-03 (Estimated); Results first posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- tDCS anodal stimulation (Experimental): anodal stimulation
  Interventions: Device: tDCS
- tDCS cathodal stimulation (Active Comparator): cathodal stimulation
  Interventions: Device: tDCS
- Sham stimulation (Sham Comparator): Sham stimulation. Termination of electrical stimulation following 30 seconds
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — comparing anodal, cathodal, and sham tDCS

SUMMARY:
This study will examine the benefits of transcranial direct current stimulation (tDCS), a new tool that is being developed as a safe and non-invasive neurostimulation method, for improving neurocognitive and social cognitive functions in schizophrenia. This procedure is non-invasive and painless and it results in increase or decrease of spontaneous neuronal firing in the brain. Its safety and beneficial effect on cognition has been demonstrated in healthy individuals and several clinical populations. In this pilot study, the investigators will examine the effect of tDCS on cognitive functions in 40 individuals with schizophrenia. Each participant will arrive for three visits, with approximately one week between each visit. During the first visit, participants will be interviewed about their psychiatric symptoms, personal life experiences, and emotional well being by a specially-trained interviewer. On each of the three visits, participants will receive one of three stimulations: a type of tDCS designed to increase neuronal firing, an alternative form of tDCS designed to decrease neuronal firing, and a sham tDCS (stimulation with no current). Immediately following the stimulation, participants will be asked to complete measures of mental abilities, including tests presented on a computer screen and paper-and-pencil tests. During each visit, participants will also undergo a standard measure of brain activity (EEG) while listening to tones. The first visit will last approximately five hours, and the other two visits will last approximately four hours each. The project will take approximately two years to complete.

DETAILED DESCRIPTION:
The investigators plan to recruit 40 individuals diagnosed with Schizophrenia. Participants will range from 18-55 years old. We will select stable, medicated patients who have not been hospitalized nor had any changes in their antipsychotic medications during the previous two months. Participants will not be tested within 12 hours of taking medications that may affect cognition (such as benzodiazepines and anticholinergics). All medications will be recorded. The investigators expect most of the patients to be relatively chronic (mean illness chronicity approximately 15 years, based on previous studies), although we will not select for chronicity.

All participants will provide written informed consent after receiving a full explanation of the procedures according to approvals by the Institutional Review Boards. They will arrive for three visits. In the first visit, they will be consented, complete the diagnostic interview, the rating scales, and will undergo one of three randomly assigned stimulation conditions: 1) anodal tDCS, 2) cathodaltDCS, and 3) sham stimulation. They will also undergo an electroencephalography (EEG) procedure, in order to more directly assess the effect of tDCS on brain function. This visit will take approximately five hours to complete, and breaks will be given as needed. Immediately following stimulation, participants will complete neurocognitive, social cognitive, and EEG measures. There will be two 20-minute stimulation sessions, with a break of one hour between the sessions. After each session, participants will be asked to complete a portion of the basic cognitive, social cognitive, and EEG measures, so that half of the measures will be completed after the first 20 minute stimulation session and the other half will be completed after the second 20 minute stimulation session. The order of administration of the neurocognitive, social cognitive, and EEG measures will be randomized across participants within each group. During the second and third visits, participants will undergo the remaining two stimulation conditions, one randomly assigned condition each visit. These visits will take approximately four hours to complete, and each visit will be separated by at least one week from the previous visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders (DSM)-V Diagnosis of Schizophrenia
* Must understand spoken English sufficiently to comprehend testing procedures
* Estimated premorbid intelligence quotient (IQ) > 70 (based on reading ability)
* Ongoing care of a Psychiatrist, Psychologist, or other qualified mental health professional

Exclusion Criteria:

* Metal in cranium
* Cardiac lines/pacemaker
* Medication pump
* Increased intracranial pressure
* Lifetime history of serious head injury (LOC > 1 hr.)
* Sedatives or Benzodiazepines within 12 hours of testing
* Clinically significant neurological disease (e.g., seizures)
* History of mental retardation or developmental disability
* Alcohol or substance dependence in the last 6 months
* Alcohol or substance abuse in the last 1 month
* Change in medication in past 6 weeks
* Change in in living situation in the last 2 months
* Inpatient hospitalization in past 3 months
* Participation in prior studies involving tDCS

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Rassovsky, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute for Neuroscience and Human Behavior, Los Angeles, California, United States

REFERENCES:
- [Derived] Rassovsky Y, Dunn W, Wynn JK, Wu AD, Iacoboni M, Hellemann G, Green MF. Single transcranial direct current stimulation in schizophrenia: Randomized, cross-over study of neurocognition, social cognition, ERPs, and side effects. PLoS One. 2018 May 7;13(5):e0197023. doi: 10.1371/journal.pone.0197023. eCollection 2018. PMID 29734347

RESULTS

PARTICIPANT FLOW:
Groups:
- Anodal Cathodal Sham: anodal stimulation, followed by cathodal stimulation, followed by sham stimulation
- Cathodal Sham Anodal: cathodal stimulation, followed by sham stimulation, followed by anodal stimulation
- Sham Anodal Cathodal: sham stimulation, followed by anodal stimulation, followed by cathodal stimulation
Period: Overall Study
Arm/Group | Anodal Cathodal Sham | Cathodal Sham Anodal | Sham Anodal Cathodal
Started | 12 | 13 | 13
Completed | 12 | 12 | 13
Not Completed | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: tDCS: comparing anodal, cathodal, and sham tDCS
Arm/Group | All Study Participants
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cognition on MCCB
Description: Summary score of the cognitive domains on the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB). Four nonsocial neurocognitive tasks were included: speed of processing, working memory, verbal memory, and reasoning/problem solving. Normed T-scores were calculated for each cognitive subdomain, as well as the cognitive composite score consisting of the average across the four subdomains. The T-scores have a mean of 50, with a difference of 10 points from the mean equaling one standard deviation. Higher T-scores are indicative of higher cognition.
Time Frame: baseline and 20 minutes
Measure: Mean (Standard Error); unit: T-scores
Groups:
- Sham Stimulation: Termination of electrical stimulation following 30 seconds
  tDCS: comparing anodal, cathodal, and sham tDCS
Arm/Group | tDCS Anodal Stimulation | tDCS Cathodal Stimulation | Sham Stimulation
Number analyzed (Participants) | 37 | 37 | 37
T-scores | 45.0 (1.65) | 45.2 (1.65) | 45.8 (1.64)

2. Primary Outcome: Change From Baseline in Managing Emotions on MSCEIT
Description: Total score on the Managing Emotions component of Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT) The test consists of 141 items and 8 ability subtests, which assess four components of emotional processing. In this study, only branches 1 and 4 were administered, focusing on the Managing Emotions component. The total score reflects mean performance across the branches. The scores were converted to normed T-scores that have a mean of 50, with a difference of 10 points from the mean equaling one standard deviation. Higher T-scores are indicative of better performance.
Time Frame: baseline and 20 minutes
Measure: Mean (Standard Error); unit: T-scores
Arm/Group | tDCS Anodal Stimulation | tDCS Cathodal Stimulation | Sham Stimulation
Number analyzed (Participants) | 37 | 37 | 37
T-scores | 36.4 (2.06) | 37.7 (2.05) | 37.1 (2.05)

ADVERSE EVENTS:
Time Frame: Following every tDCS administration
Description: Standard questionnaire.
Arm/Group | tDCS Anodal Stimulation | tDCS Cathodal Stimulation | Sham Stimulation
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37 | 0/37

LIMITATIONS AND CAVEATS:
The present findings employed a single tDCS administration, which may be insufficient to attain potential therapeutic effects. These findings thus add to the growing body of evidence suggesting the need for basic dose-finding studies in tDCS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No